CLINICAL TRIAL: NCT02419833
Title: Randomized Study of ImmeDiate Versus DeLayEd Invasive Intervention in Patients With Non ST-segment Elevation Myocardial Infarction
Brief Title: Immediate Versus Delayed Invasive Intervention for Non-STEMI Patients
Acronym: RIDDLE-NSTEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Aleksandra Milosevic, MD, Clinical Centre of Serbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 440/VII/1
Record Dates: First submitted 2015-03-09; First posted 2015-04-17 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Myocardial Infarction
Keywords: non-STEMI; immediate; delayed; PCI
MeSH Terms: conditions — Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate invasive intervention (Experimental): Invasive coronary angiography followed by either percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) surgery as soon as possible and/or within 2 hours of admission
  Interventions: Procedure: Immediate invasive intervention; Device: Coronary artery stenting
- Delayed invasive intervention (Active Comparator): Invasive coronary angiography followed by either percutaneous coronary intervention (PCI) and/or coronary artery bypass graft (CABG) surgery during the hospitalization and within 2-72 hours of admission
  Interventions: Procedure: Delayed invasive intervention; Device: Coronary artery stenting

INTERVENTIONS:
Procedure: Immediate invasive intervention — Invasive coronary angiography followed by either percutaneous coronary intervention (PCI) and/or coronary artery bypass graft (CABG) surgery as soon as possible and/or within 2 hours of admission
  Arms: Immediate invasive intervention
Procedure: Delayed invasive intervention — Invasive coronary angiography followed by either percutaneous coronary intervention (PCI) and/or coronary artery bypass graft (CABG) surgery during the hospitalization and/or within 2-72 hours of admission
  Arms: Delayed invasive intervention
Device: Coronary artery stenting — Implantation of coronary stents

SUMMARY:
In patients with acute myocardial infarction without ST-segment elevation on ECG (non-STEMI), previous studies have indicated that routine invasive treatment confers more benefit as compared to selective invasive approach. The benefits of routine invasive coronary intervention have been the most evident in patients with higher baseline risk profile. However, the question of optimal timing of routine invasive intervention remains unsolved.

Immediate invasive intervention early after admission for non-STEMI may limit myocardial necrosis by securing the patency of the culprit coronary artery. Nevertheless, several previous studies reported higher levels of biomarkers of myocardial injury in patients undergoing early PCI. The question of earlier versus delayed procedure in non-STEMI patients may thus amount to whether the risk of intervening on an unstable plaque is greater than the risk of new ischemic events while waiting for the invasive procedure.

The purpose of the present study is to compare effects of immediate coronary intervention, within 2 hours of admission, versus delayed intervention, within 2-72 hours after admission, in patients witn non-STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. episode of chest pain occurring no longer than 24 hours prior to admission
2. elevation of cardiac troponin I above the upper limit of normal (ULN)
3. new ST-segment depression at least 1 millivolt (mV) and/or T-wave inversion or transient ST-segment elevation in ≥ 2 contiguous leads

Exclusion Criteria:

1. age < 18 years
2. persistent ST-segment elevation
3. hemodynamic instability
4. cardiogenic shock on admission
5. life-threatening ventricular arrhythmias on admission
6. refractory angina on admission
7. active bleeding
8. any contraindication for the use of dual antiplatelet therapy (DAPT)
9. presence of comorbidities with life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2009-09; Primary Completion 2013-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause death or myocardial reinfarction | within 30 days of randomization

SECONDARY OUTCOMES:
Composite of all-cause death, myocardial reinfarction or recurrent ischemia | within 30 days of randomization
All-cause mortality | within 30 days, 1, 3 and 5 years after randomization
Myocardial reinfarction | within 30 days, 1, 3 and 5 years after randomization
Stroke | within 30 days, 1, 3 and 5 years after randomization
Recurrent ischemia | within 30 days of randomization
Major bleeding | within 30 days, 1, 3 and 5 years after randomization
Duration of index hospitalization | at 30-day follow-up, the duration of hospital stay is assessed

CONTACTS AND LOCATIONS:
Overall Officials: Goran Stankovic, MD, PhD, Study Director — Clinical Centre of Serbia; Aleksandra Milosevic, MD, Principal Investigator — Clinical Centre of Serbia; Zorana Vasiljevic, MD, PhD, Study Chair — Clinical Centre of Serbia
Locations (1):
- Clinical Centre of Serbia, Department of Cardiology, Belgrade, Serbia

REFERENCES:
- [Derived] Milosevic A, Vasiljevic-Pokrajcic Z, Milasinovic D, Marinkovic J, Vukcevic V, Stefanovic B, Asanin M, Dikic M, Stankovic S, Stankovic G. Immediate Versus Delayed Invasive Intervention for Non-STEMI Patients: The RIDDLE-NSTEMI Study. JACC Cardiovasc Interv. 2016 Mar 28;9(6):541-9. doi: 10.1016/j.jcin.2015.11.018. Epub 2016 Jan 6. PMID 26777321